CLINICAL TRIAL: NCT04656483
Title: Supporting Parenting at Home: Empowering Rehabilitation Through Engagement (SPHERE)
Acronym: SPHERE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SPHERE
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Neurodevelopmental Disorders
Keywords: early family-centered intervention; telemedicine; video feedback; parenting; telerehabilitation; disability; psychomotor delay
MeSH Terms: conditions — Neurodevelopmental Disorders; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Video Feedback Arm (Experimental): Mother-child dyads will take part into a 6 video-conference sessions of Video Feedback (vVF). The vVF will be standardized according to previously published RCTs. Specifically, the 6 vVFI sessions will be organized in two subsequent phases: 4 sessions based on sharing the focus on different relational themes, and 2 sessions of interactive integration. In more specific terms, during the first set of 4 sessions the psychologist will review with mothers' segments of the videotapes obtained during the baseline assessment and will focus on four different relational themes: responsiveness, physical stimulation, teaching, and parenting experience. During the interactive integration session, the insights developed from the first 4 videoconferences will be applied to the real-time interaction between the parent and his/her infant under the guidance of the psychologist.
  Interventions: Other: Telemedicine Video Feedback Intervention
- Psychoeducational booklet arm (Active Comparator): Mothers assigned to condition B will receive an informative booklet addressing the same themes discussed in the experimental intervention (i.e., responsiveness, physical stimulation, teaching, and parenting experience), but not tailored on their own infant or specific parenting challenges.
  Interventions: Other: Psychoeducational Booklet Intervention

INTERVENTIONS:
Other: Telemedicine Video Feedback Intervention — Mother-child dyads will take part into a 6 video-conference sessions of Video Feedback (vVF). The vVF will be standardized according to previously published RCTs. Specifically, the 6 vVFI sessions will be organized in two subsequent phases: 4 sessions based on sharing the focus on different relational themes, and 2 sessions of interactive integration. In more specific terms, during the first set of 4 sessions the psychologist will review with mothers' segments of the videotapes obtained during the baseline assessment and will focus on four different relational themes: responsiveness, physical stimulation, teaching, and parenting experience. During the interactive integration session, the insights developed from the first 4 videoconferences will be applied to the real-time interaction between the parent and his/her infant under the guidance of the psychologist.
  Arms: Telemedicine Video Feedback Arm
Other: Psychoeducational Booklet Intervention — Mothers of this condition will receive an informative booklet addressing the same themes included in the experimental intervention (responsiveness, physical stimulation, teaching, and parenting experience), but not tailored on their own infant status.
  Arms: Psychoeducational booklet arm

SUMMARY:
Infants with Neurodevelopmental Disabilities (ND) show emotional, cognitive and socio-interactive dysregulation dramatically impacting on caregiving behavior. Early family-centered rehabilitation interventions are effective in promoting better infant outcomes and in optimizing healthcare systems economic return in the long-term. The Video Feedback intervention (VFI) is effective in promoting sensitive parenting and supporting infants' development. In the light of limited resources of the healthcare systems, technological advance in telemedicine may facilitate the delivery of VFI to a greater number of families of infants with ND. Consistently, the Supporting Parenting at Home: Empowering Rehabilitation through Engagement (SPHERE) project is a randomized controlled trial (RCT) aiming at assessing effectiveness and efficacy of an early family centered VFI parenting support delivered through videoconferencing on dyads with infants with ND.

DETAILED DESCRIPTION:
Infants with Neurodevelopmental Disabilities (ND) show emotional, cognitive and socio-interactive dysregulation dramatically impacting on caregiving behavior. Parents may report critical emotional burden with heightened risk for chronic levels of distress, depression and anxiety. This constitutes a crucial point considering that parenting represents the first preventive factors for infants' development also in the presence of ND conditions. Thus, it is not surprising that early rehabilitation interventions that focus on the parent-infant dyad have been found to be the most effective in recent meta-analytic study and to be the most rewarding for healthcare systems in terms of economic return in the long-term. Specifically, the VFI constitutes an early family-centered intervention that proved to be effective in promoting sensitive parenting and supporting infants' behavioral and socio-emotional development. The use of VFI intervention has been also documented to be beneficial in dyads of children with neurodevelopmental disability reducing child's disruptive and emotionally negative behaviors; promoting maternal sensitivity, increasing self- efficacy and reducing parenting stress. It should be highlighted that delivering VFI in hospital or home-based context should be highly demanding for the healthcare systems due to high cost and disparities in access to the service for families in remote areas. As such, delivering VFI through telemedicine approaches (e.g., videoconferencing) appears to hold promises of promoting a reduction in inequality of care, greater access to early family-centered support and a more effective and efficient promotion of health outcomes for infants with ND. We still do not know how a VFI support for parents of infants with ND may end up in being effective and efficient in terms of promoting infants' development and parental health. Consistently, the Supporting Parenting at Home: Empowering Rehabilitation through Engagement (SPHERE) project is a randomized controlled trial (RCT) aiming at assessing effectiveness of an early family centered VFI parenting support delivered through videoconferencing on dyads with infants with ND.

The SPHERE RCT will include two arms (see arm description) and three assessment phases: T0, baseline; T1, immediate post-intervention; T2, follow-up (6 months after the intervention). For both arms, standardized assessment sessions will include video-recording of mother-infant interaction and maternal self-report scales (depression [Beck Depression Inventory, BDI; Beck et al., 1961]; anxiety [State-Trait Anxiety Inventory, STAI-Y, Spielberg, 1983] parenting stress, [Parenting Stress Index, PSI; Abidin, 1983] and infants' temperament [Infant Behavior Questionnaire Revised, IBQ-R, Gartstein et al., 2003]).

ELIGIBILITY:
Inclusion Criteria:

* infants' (corrected) age between 1 and 18 months;
* presence of developmental risk or diagnosis of ND as defined by standardized clinical criteria;
* parental age greater than 18 years;
* parental mastery of Italian language;
* parents living together with the infant.

Exclusion Criteria:

* Twins;
* Infant's life-threatening conditions;
* Maternal full-blown documented psychiatric disorders.

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity | Immediate post-intervention (6 weeks after the intervention started)
  The maternal sensitivity will be coded through the Global Rating Scales (Murray, Fiori-Cowley, Hooper, & Cooper, 1996). The score will range from 1 (low) to 5 (high).

SECONDARY OUTCOMES:
Infant emotional stress reactivity | Immediate post-intervention (6 weeks after the intervention started)
  It will be coded as infant negative emotionality through the infant's emotionality coding system (Brambilla et al., 2020; unpublished manual). The proportion of time in which the infant will be positive, neutral or negative will be obtained (score range for each emotion: 0 to 1).
Maternal sensitivity | Follow-up (6 months adfter the intervention ended)
  The maternal sensitivity will be coded through the Global Rating Scales (Murray, Fiori-Cowley, Hooper, & Cooper, 1996). The score will range from 1 (low) to 5 (high).
Infant emotional stress reactivity | Follow-up (6 months adfter the intervention ended)
  It will be coded as infant negative emotionality through the infant's emotionality coding system (Brambilla et al., 2020; unpublished manual). The proportion of time in which the infant will be positive, neutral or negative will be obtained (score range for each emotion: 0 to 1).

OTHER OUTCOMES:
Maternal Stress | Immediate post-intervention (6 weeks after the intervention started)
  Measured through the self-report scale Parenting Stress Index (PSI; Abidin, 1983). PSI total score ranges from 36 (low) to 180 (high).
Maternal Stress | Follow-up (6 months adfter the intervention ended)
  Measured through the self-report scale Parenting Stress Index (PSI; Abidin, 1983). PSI total score ranges from 36 (low) to 180 (high).
Maternal depression | Immediate post-intervention (6 weeks after the intervention started)
  Measured through the self-report Beck Depression Inventory (BDI; Beck et al, 1988). BDI total score ranges from 0 (low) to 63 (high).
Maternal depression | Follow-up (6 months adfter the intervention ended)
  Measured through the self-report Beck Depression Inventory (BDI; Beck et al, 1988). BDI total score ranges from 0 (low) to 63 (high).
Maternal anxiety | Immediate post-intervention (6 weeks after the intervention started)
  Measured through the state subscale of the self-report State-Trait Anxiety Inventory (STAI; Spielberger et al., 1983). The state subscale score ranges from 20 (low) to 80 (high).
Maternal anxiety | Follow-up (6 months adfter the intervention ended)
  Measured through the state subscale of the self-report State-Trait Anxiety Inventory (STAI; Spielberger et al., 1983). The state subscale score ranges from 20 (low) to 80 (high).
Infant temperament regulation | Immediate post-intervention (6 weeks after the intervention started)
  Measured through the mother-report Infant Behavior Questionnaire-Revised (Gartstein & Rothbart, 2003). The IBQ-R subscale of interest is the "Orienting/Regulatory Capacity". Its score ranges from 1 (low) to 7 (high).
Infant temperament regulation | Follow-up (6 months adfter the intervention ended)
  Measured through the mother-report Infant Behavior Questionnaire-Revised (Gartstein & Rothbart, 2003). The IBQ-R subscale of interest is the "Orienting/Regulatory Capacity". Its score ranges from 1 (low) to 7 (high).

CONTACTS AND LOCATIONS:
Overall Officials: Serena Grumi, PhD, Principal Investigator — IRCCS Mondino Foundation, Pavia, Italy; Livio Provenzi, PhD, Study Chair — IRCCS Mondino Foundation, Pavia, Italy
Locations (1):
- Mondino Foundation, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grumi S, Borgatti R, Provenzi L. Supporting Parenting at Home-Empowering Rehabilitation through Engagement (SPHERE): study protocol for a randomised control trial. BMJ Open. 2021 Dec 14;11(12):e051817. doi: 10.1136/bmjopen-2021-051817. PMID 34907057